CLINICAL TRIAL: NCT00776191
Title: Randomized, Multicenter Cross-over Study in Investigating the Effect of Bicarbonate-based Solutions (Physioneal 35 vs. 40) on Protein Metabolism in Children and Adolescents on Chronic Peritoneal Dialysis
Brief Title: Randomized Multicenter Cross-over Study to Compare the Effect of Physioneal 35 to 40 on the Protein Metabolism
Acronym: NephropaedPD01
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: al study sites stoped on 15/05/2012 because of insufficient recrutement.
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2005-005434-12
Record Dates: First submitted 2008-10-20; First posted 2008-10-21 (Estimated); Last update posted 2015-06-04 (Estimated); Status verified 2015-06

CONDITIONS: Endstage Renal Disease
Keywords: Physioneal 35; Physioneal 40; children; chronic peritoneal dialysis
MeSH Terms: interventions — Physioneal 35; Physioneal 40

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Physioneal 35 vs. 40 (Active Comparator): Physioneal 35® Glucose solution with Bicarbonate 25 mmol/l, Lactate 10 mmol/l, and Calcium 1.75 mmol/l for eight weeks, followed by Physioneal 40® Glucose solution Bicarbonate 25 mmol/l, Lactate 15 mmol/l, and Calcium 1.25 mmol/l for eight weeks.
  Interventions: Drug: Physioneal 35
- Physioneal 40 vs. 35 (Active Comparator): Physioneal 40® Glucose solution Bicarbonate 25 mmol/l, Lactate 15 mmol/l, and Calcium 1.25 mmol/l for eight weeks followed by Physioneal 35® Glucose solution with Bicarbonate 25 mmol/l, Lactate 10 mmol/l, and Calcium 1.75 mmol/l for eight weeks
  Interventions: Drug: Physioneal 40

INTERVENTIONS:
Drug: Physioneal 35 — Physioneal 35® for eight weeks, followed by Physioneal 40® for eight weeks
  Other Names: Nephropaed-PD-01/B
  Arms: Physioneal 35 vs. 40
Drug: Physioneal 40 — Physioneal 40® for eight weeks followed by Physioneal 35® for eight weeks
  Other Names: Nephropaed-PD-01/B
  Arms: Physioneal 40 vs. 35

SUMMARY:
The purpose of this study is to demonstrate an increase in protein metabolism during treatment with Physioneal 35® (containing lactate 10 mmol/l, calcium 1.75 mmol/l) compared to treatment with Physioneal 40® (containing lactate 15 mmol/l, calcium 1.25 mmol/l) in children and adolescents with end stage renal failure receiving peritoneal dialysis.

DETAILED DESCRIPTION:
* Fat oxidation (13C-enrichment in expiration breath samples for U-C13-algae turnover)
* Growth markers (plasma levels of IgF-1, IgF-BP3, leptin)
* Biochemical markers of anabolism (plasma levels of total protein, albumin, transferrin)
* Serum thyroid function (fT3, fT4, TSH)
* Serum lipid status
* Serum markers of calcium/phosphate metabolism (PTH, calcium, ionized calcium, phosphate, alkaline phosphatase)
* Prevalence of metabolic acidosis/ alkalosis (venous sample), serum lactate
* Safety parameters (such as normalized weekly Kt/v, parameters of glucose metabolism, parameters of hepatic function, parameters of calcium-phosphate-metabolism, physical examination incl. standing height, weight, assessment of complications related to peritoneal dialysis as peritonitis, exit infections and inguinal hernia)
* Body composition (lean body mass and body fat mass/fluid)

ELIGIBILITY:
Inclusion Criteria:

* Patients who are males or non-pregnant females between the ages of 3 months and 18 years.
* Patients who are on regular automated peritoneal dialysis due to end stage renal failure for at least 3 months.
* Patients and/or their parents must be capable of understanding the purpose and risks of the study.
* Patients and/or their parents (or guardians) who are willing to give written informed consent and willing to participate in and comply with the study protocol.

Exclusion Criteria:

* Use of pure lactate, amino acid or oligosaccharide solutions for peritoneal dialysis
* Peritonitis episode less than 6 weeks before enrolment
* Hypercalcemia (serum) > 2.75 mmol/l in three independent measurements during 10 days
* Severe secondary hyperthyroidism (iPTH > 500 ng/l)
* Renal anemia with hemoglobin (blood) < 10 mg/dl
* Impaired hepatic function (AST/SGOT or ALT/SGPT > 2 times the upper limit of the reference range)
* Patients who are participating in another study that requires Ethics Committee approval. Non-interventional studies are permitted.
* Pregnant female patients, females of childbearing potential who are unwilling or unable to use adequate contraception methods.
* Severe respiratory insufficiency
* Malnourishment (body weight < -2.5 SDS for height and gender) or severe deterioration of fat metabolism
* Patients with a history of malignancy of any organ system, treated or untreated
* Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism, or excretion of the investigational product and the comparator, including

  * Major deterioration of the abdominal wall (e.g. dermal infections or burns, hernia)
  * Major deterioration of the abdominal cavity (e.g. ascites, ileus, adhesions, bowel perforation, defects of the diaphragm, tumours)
* Patients with a history of viral infections such as HIV or hepatitis B, C.

Ages: 3 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Actual)
Dates: Start 2008-09; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
To demonstrate an increase in protein metabolism during treatment with Physioneal 35® compared to treatment with Physioneal 40® in children and adolescents with end stage renal failure receiving peritoneal dialysis. | 16 weeks

SECONDARY OUTCOMES:
To demonstrate a improved Fat oxidation during treatment with Physioneal compared to treatment with Physioneal 40® in children and adolescents with end stage renal failure receiving peritoneal dialysis. | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Joerg Doetsch, Prof. Dr., Principal Investigator — University Hospital Erlangen, Department of Pediatrics University Hospital Koeln
Locations (5):
- Germany (5):
  - Pediatric Nephrology, Universiy Children's Hospital, Cologne
  - Dept. of Pediatric Nephrology, University Hospital Erlangen, Erlangen
  - Dept. of Pediatric Nephrology, University of Hannover, Hanover
  - Dept. of Nephrology, children´s hospital Memmingen, Memmingen
  - Dept. of Nephrology, University of Rostock, Rostock